CLINICAL TRIAL: NCT03672435
Title: Does Proparacaine Enhance Strabismus Recovery
Brief Title: Strabismus Recovery With Proparacaine and Oculocardiac Reflex
Acronym: OCRprop
Status: Completed | Type: Observational
Sponsor: Alaska Blind Child Discovery (Other)
Responsible Party: Sponsor
Other Study IDs: ABCD OCR proparacaine
Record Dates: First submitted 2018-09-06; First posted 2018-09-14 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2018-09

CONDITIONS: Strabismus; Bradycardia; Nausea; Pain
Keywords: post operative recovery; oculocardiac reflex; extra ocular muscle; conjunctiva; numbing drop; heart rate
MeSH Terms: conditions — Strabismus; Bradycardia; Nausea; Pain | interventions — Solutions; proxymetacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- proparacaine: Received topical proparacaine 0.5% with routine antibiotic-steroid ointment in operative eye(s) following strabismus surgery
  Interventions: Drug: Topical Solution
- No proparacaine: Received no topical proparacaine 0.5% but did receive routine antibiotic-steroid ointment in the operative eye(s) following strabismus surgery

INTERVENTIONS:
Drug: Topical Solution — proparacaine 0.5% eye drop
  Other Names: proparacaine
  Groups: proparacaine

SUMMARY:
Observational study to determine if topical anesthetic and intraoperative oculocardiac reflex influence post strabismus surgery recovery.

DETAILED DESCRIPTION:
In an observational study with de-identified data of oculocardiac reflex (OCR) and strabismus surgery under routine anesthesia, a cohort of ongoing patients received topical proparacaine immediately post op, or none. Co-variables were intraoperative opioid and OCR, patient age, type of surgery. Several post-operative recovery outcome variables were prospectively monitored.

ELIGIBILITY:
Inclusion Criteria:

* Strabismus surgery

Exclusion Criteria:

* none

Ages: 3 Months to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: strabismus surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2010-07-29 (Actual); Primary Completion 2013-11-21 (Actual); Study Completion 2013-11-21 (Actual)

PRIMARY OUTCOMES:
pain (post op pain Likert scale) | hours (1-4) in recovery room
  pain scale description / observation.. Pain is ranked by patient or nurse from 0 (no pain) to 9 (much pain)

SECONDARY OUTCOMES:
nausea | hours (1-4) in recovery room
  observed or described nausea (presence or absence of nausea / vomiting)
heart rate | hours (1-4) while in recovery room
  recovery room heart rate
time to recovery | minutes (30-240) from entry recovery room to discharge
  time in recovery room

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Arnold, MD, Principal Investigator — Alaska Blind Child Discovery

IPD SHARING:
Plan to Share IPD: Yes
Study Website access
Supporting Information: Study Protocol
Time Frame: current- ongoing
Access Criteria: public
URL: http://www.abcd-vision.org/OCR/index.html

REFERENCES:
- [Background] Arnold RW, Bond AN. Does Topical Proparacaine Improve Postoperative Comfort After Strabismus Surgery? Clin Ophthalmol. 2019 Nov 20;13:2279-2283. doi: 10.2147/OPTH.S230498. eCollection 2019. PMID 31819352
- [Result] Arnold RW, Biggs RE, Beerle BJ. Intravenous dexmedetomidine augments the oculocardiac reflex. J AAPOS. 2018 Jun;22(3):211-213.e1. doi: 10.1016/j.jaapos.2018.01.016. Epub 2018 May 5. PMID 29733898
- Available data/document: Individual Participant Data Set — http://www.abcd-vision.org/OCR/OCR%20proparacaine%20de-identified.pdf — deidentified OCR topical anesthetic recovery outcomes